CLINICAL TRIAL: NCT03251469
Title: Single Dose of Tranexamic Acid at the Time of Surgery and Blood Loss, in Elderly Patients Undergoing Hip Fracture Surgery
Brief Title: Single Dose of Tranexamic Acid and Blood Loss, in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vasileios S. Nikolaou, Assistant Professor of Orthopaedics, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2016-11-29; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Blood Loss, Surgical; Hip Fractures; Complication, Postoperative
Keywords: tranexamic acid; blood tranfusion; hip fractures; elderly; blood loss
MeSH Terms: conditions — Blood Loss, Surgical; Hip Fractures; Postoperative Complications; Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): intravenous tranexamic acid, 15mg/kg, preoperatively, single dose
  Interventions: Drug: Tranexamic Acid 15mg/kg , iv, Single Dose
- Group 2 (Placebo Comparator): Intravenous normal saline, 100mg, preoperatively, single dose
  Interventions: Drug: Normal Saline, 100mg, iv, Singe dose

INTERVENTIONS:
Drug: Tranexamic Acid 15mg/kg , iv, Single Dose — Tranexamic Acid 15mg/kg , administered intravenously, preoperatively, in a single dose
  Arms: Group 1
Drug: Normal Saline, 100mg, iv, Singe dose — Normal Saline, 100mg, administered intravenously, preoperatively in single dose
  Arms: Group 2

SUMMARY:
The aim of this study is to investigate the hypothesis that single dose of tranexamic acid (TXA) preoperatively will lower blood loss and transfusion rate in elderly patients with hip fractures (intertrochanteric or Subcapital), that will be treated with intramedullary nailing and cemented hemiarthroplasty respectively. After application of inclusion and exclusion criteria, patients will be randomized in two groups. Group 1 will include patients that receive preoperatively single dose of TXA (15mg/kg) and Group 2 will include patients that receive normal saline (control group).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive elderly patients (age >75 yo) undergoing hip fracture surgery for a stable or unstable intertrochanteric hip fracture with the insertion of a short intramedullary nail (IMN) as well as patients treated surgically with cemented hemiarthroplasty for acute femoral neck (subcapital) hip fracture.

Exclusion Criteria:

* Any contraindication for tranexamic acid
* Multiple fractures
* Requirement for anticoagulant therapy that could not be stopped.
* Ongoing thromboembolic event
* reduced kidney function
* malignancy,
* pathological fracture
* previous operation on the affected hip
* Active coronary artery disease (event in the past 12 months).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
number of transfusions of allogeneic RBC from surgery up to day 4 | 5 days
total blood loss from surgery to day | 5 days

SECONDARY OUTCOMES:
incidence of vascular events | 3 months
Incidence of deaths | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Orthopaedics, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No